CLINICAL TRIAL: NCT05934591
Title: Improving Attendance in Community Wise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Comprehensive Behavioral Health Center (Unknown)
Responsible Party: Principal Investigator, Liliane Cambraia Windsor, Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: UIUC IRB 23828
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Results first posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Intervention Engagement and Retention
Keywords: Alcohol and substance misuse treatment, treatment engagement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Supervision/Paid/Open Group (Experimental): A group of people under supervision (those on parole, drug court, probation, or methadone maintenance) will receive an incentive to attend open format groups of the Community Wise intervention.
  Interventions: Behavioral: Community Wise
- Supervison/Paid/Closed Group (Experimental): A group of people under supervision (those on parole, drug court, probation, or methadone maintenance) will receive an incentive to attend closed format groups of the Community Wise intervention.
  Interventions: Behavioral: Community Wise
- Supervision/Not Paid/Open Group (Experimental): A group of people under supervision (those on parole, drug court, probation, or methadone maintenance) will attend open format groups of the Community Wise intervention without receiving an incentive.
  Interventions: Behavioral: Community Wise
- Supervision/Not Paid/Closed Group (Experimental): A group of people under supervision (those on parole, drug court, probation, or methadone maintenance) will attend closed format groups of the Community Wise intervention without receiving an incentive.
  Interventions: Behavioral: Community Wise
- Not Under Supervision/Paid/Open Group (Experimental): A group of people not under supervision (those on parole, drug court, probation, or methadone maintenance) will receive an incentive to attend open format groups of the Community Wise intervention.
  Interventions: Behavioral: Community Wise
- Not Under Supervision/Paid/Closed Group (Experimental): A group of people not under supervision (those on parole, drug court, probation, or methadone maintenance) will receive an incentive to attend closed format groups of the Community Wise intervention.
  Interventions: Behavioral: Community Wise
- Not Under Supervision/Not Paid/Open Group (Experimental): A group of people not under supervision (those on parole, drug court, probation, or methadone maintenance) will attend open format groups of the Community Wise intervention without receiving an incentive.
  Interventions: Behavioral: Community Wise
- Not Under Supervision/Not Paid/Closed Group (Experimental): A group of people not under supervision (those on parole, drug court, probation, or methadone maintenance) will attend closed format groups of the Community Wise intervention without receiving an incentive.
  Interventions: Behavioral: Community Wise

INTERVENTIONS:
Behavioral: Community Wise — The intervention received by each group will be Community Wise, a multi-level manualized behavioral intervention to decrease alcohol and substance misuse frequency

SUMMARY:
Rates of alcohol and substance misuse (ASM) in low-income, predominantly African American communities are similar to the general population. However, ASM has greater consequences (e.g., higher incarceration and HIV infection rates) for residents in these communities. We developed and optimized Community Wise (CW), a multi-level manualized behavioral intervention to decrease ASM frequency in a population of self-identified men with histories of substance use disorder (SUD) and incarceration (SUD) in Essex County, New Jersey (NJ), U.S. We propose a study to: 1) identify strategies to improve attendance and reduce ASM, and 2) to test feasibility and acceptability of CW among self-identified men and women with a history of SUD living in marginalized communities. We will achieve these aims by conducting a 23 full factorial experiment informed by MOST and CBPR. This study will identify efficient, scalable, and sustainable strategies to improve attendance and hence, maximize the interventions' effect in reducing ASM.

DETAILED DESCRIPTION:
Rates of alcohol and substance misuse (ASM) in low-income, predominantly African American communities (from here on marginalized communities) are similar to the general population. However, ASM has greater consequences (e.g., higher incarceration and HIV/HCV infection rates) for residents in these communities. While the etiology underpinning this inequity is complex, the root cause of these issues has been traced to social determinants of health (SDH; e.g., stigma; poverty; barriers to education, housing, and employment).

Funded by the National Institute for Minority Health Disparities (NIMHD 5R01MD010629), in partnership with the Critical Consciousness Collaborative Board (3CB), we developed Community Wise (CW), a multi-level manualized behavioral intervention to decrease ASM frequency in a population of self-identified men with histories of substance use disorder (SUD) and incarceration in Essex County, NJ, U.S. The 3CB was founded in 2010 and developed and pilot-tested the original CW. Over the past six years, our team used the multiphase optimization strategy (MOST), and community based participatory research (CBPR) principles to develop and optimize CW for efficacy in reducing ASM and cost. MOST is an innovative methodological framework that employs experimental designs to engineer efficient and effective behavioral interventions. MOST guided the optimization of CW with delivery cost of less than $2,000 per intervention cycle serving up to ten individuals simultaneously (this was the Medicaid allowable reimbursement cost for SUD group treatment services in 2015). Clinical trial results showed larger ASM reduction (Cohen's d=-2∙22, P=0∙067) in the optimized CW group. Unfortunately, attendance across the 15 intervention sessions was low (only 15% of participants attended 50% of the sessions). Low attendance was due to the intervention's closed group format, the study's randomization strategy, and instability of the study's population (homelessness, poverty).

In order to improve upon our positive results and maximize our chances to successfully obtain further external funding to test CW effectiveness, we need funding to: 1) identify strategies to improve attendance and reduce ASM, and 2) to test feasibility and acceptability of CW among men and women with a history of SUD living in marginalized communities. We will achieve these aims by conducting a 23 full factorial experiment. This study will help us identify efficient strategies for improving attendance and, hence, maximize the interventions' effect in reducing ASM. As a highly efficient experimental design, a full factorial experiment will maximize study power and allow us to examine the individual and interactive contributions of each intervention delivery strategy on intervention attendance. MOST will inform which strategies will be retained, thus minimizing waste of resources. The current proposed research will also be conducted in partnership with the 3CB. As our primary individual level outcome, we will use number of sessions attended to test if different intervention delivery strategies will result in a clinically and statistically important intervention attendance with a minimum of 50% of participants attending at least 50% of the intervention. We will also compare the effect of different strategies on reducing ASM. Intervention delivery strategies include: 1) Recruiting individuals under supervision (those on parole, drug court, probation, or methadone maintenance); 2) Incentivizing intervention attendance; and 3) Delivering the intervention in an open group format. We will also compare intervention satisfaction measures between intervention strategies.

We will expand eligibility criteria to include women and people with SUD living in marginalized communities who have not been previously incarcerated. While women comprise a smaller percentage of people with SUD, they experience significant barriers to SUD treatment. Our pilot study showed that women started the CW intervention with worse outcomes when compared to men but had significantly higher reductions of ASM. While the original CW intervention was developed with and for formerly incarcerated people, it addresses concepts that are relevant to all people with SUD living in marginalized communities. Hence, the 3CB has recommended that we expand our eligibility criteria to reach a more diverse group of people. Our 23 full factorial design will examine change in attendance (N=144). Data will be collected at baseline and three months post-baseline. This study will impact public health as it will improve the potency of an optimized multi-level intervention adaptable to address different health inequities.

ELIGIBILITY:
Inclusion Criteria:

* Living in St. Clair County, Illinois (IL)
* Over 18
* English- speaker
* Under supervision (parole, probation, drug court or methadone maintenance)
* Having an alcohol or substance misuse disorder

Exclusion Criteria:

* Not living in St. Clair County, IL
* Not able to speak English
* Not able or willing to provide consent
* Not having an alcohol or substance misuse disorder
* Under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Each of the 8 arms will include both men and women
Enrollment: 166 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Comprehensive Behavioral Health Center, East Saint Louis, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Supervision/Paid/Open Group: People under supervision (those on parole, drug court, probation, or methadone maintenance) will receive an incentive to attend open format groups of the Community Wise intervention.
- Supervision/Paid/Closed Group: People under supervision (those on parole, drug court, probation, or methadone maintenance) will receive an incentive to attend closed format groups of the Community Wise intervention.
- Supervision/Not Paid/Open Group: People under supervision (those on parole, drug court, probation, or methadone maintenance) will attend open groups of the Community Wise intervention without an incentive.
- Supervision/Not Paid/Closed Group: People under supervision (those on parole, drug court, probation, or methadone maintenance) will attend closed groups of the Community Wise intervention without an incentive.
- Not Under Supervision/Paid/Open Group: People not under supervision (those on parole, drug court, probation, or methadone maintenance) will receive an incentive to attend open groups of the Community Wise intervention.
- Not Under Supervision/Paid/Closed Group: People not under supervision (those on parole, drug court, probation, or methadone maintenance) will receive an incentive to attend closed groups of the Community Wise intervention.
- Not Under Supervision/Not Paid/Open Group: People not under supervision (those on parole, drug court, probation, or methadone maintenance) will attend open groups of the Community Wise intervention without receiving an incentive.
- Not Under Supervision/Not Paid/Closed Group: People not under supervision (those on parole, drug court, probation, or methadone maintenance) will attend closed groups of the Community Wise intervention without receiving an incentive.
Period: Overall Study
Arm/Group | Supervision/Paid/Open Group | Supervision/Paid/Closed Group | Supervision/Not Paid/Open Group | Supervision/Not Paid/Closed Group | Not Under Supervision/Paid/Open Group | Not Under Supervision/Paid/Closed Group | Not Under Supervision/Not Paid/Open Group | Not Under Supervision/Not Paid/Closed Group
Started | 15 | 20 | 25 | 22 | 32 | 22 | 15 | 15
Completed | 15 | 20 | 23 | 22 | 31 | 22 | 12 | 15
Not Completed | 0 | 0 | 2 | 0 | 1 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Not Under Supervision/Not Paid/Closed Group: People not under supervision (those on parole, drug court, probation, or methadone maintenance) will attend closed groups of the Community Wise intervention without receiving an incentive.
  Period Title: Overall Study
- Total: Total of all reporting groups
Arm/Group | Supervision/Paid/Open Group | Supervision/Paid/Closed Group | Supervision/Not Paid/Open Group | Supervision/Not Paid/Closed Group | Not Under Supervision/Paid/Open Group | Not Under Supervision/Paid/Closed Group | Not Under Supervision/Not Paid/Open Group | Not Under Supervision/Not Paid/Closed Group | Total
Number analyzed (Participants) | 15 | 20 | 25 | 22 | 32 | 22 | 15 | 15 | 166
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 20 | 25 | 21 | 32 | 21 | 14 | 14 | 162
  >=65 years | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 5 | 12 | 5 | 7 | 5 | 5 | 49
  Male | 10 | 15 | 20 | 10 | 27 | 15 | 10 | 10 | 117
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/Caribbean | 5 | 6 | 9 | 3 | 3 | 5 | 5 | 6 | 42
  African American | 6 | 5 | 4 | 5 | 21 | 12 | 5 | 5 | 63
  White | 4 | 7 | 11 | 13 | 6 | 3 | 4 | 4 | 52
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Alaskan/Native American | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3
  Other | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Missing | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 15 | 20 | 25 | 22 | 32 | 22 | 15 | 15 | 166

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Attending at Least 50% of Sessions
Description: We will test if different intervention delivery strategies will result in a clinically and statistically important intervention attendance with a minimum of 50% of participants attending at least 50% of the intervention
Time Frame: nine weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Supervision/Paid/Open Group | Supervision/Paid/Closed Group | Supervision/Not Paid/Open Group | Supervision/Not Paid/Closed Group | Not Under Supervision/Paid/Open Group | Not Under Supervision/Paid/Closed Group | Not Under Supervision/Not Paid/Open Group | Not Under Supervision/Not Paid/Closed Group
Number analyzed (Participants) | 15 | 20 | 25 | 22 | 32 | 22 | 15 | 15
Participants | 8 | 6 | 1 | 4 | 19 | 12 | 5 | 4

ADVERSE EVENTS:
Time Frame: 6 months
Description: In addition to the clinicaltrials.gov definition of an adverse event, the University of Illinois Urbana Champaign's definition of an adverse event includes "Any experience or abnormal finding that has taken place during the course of a research project and was harmful to the subject participating in the research, or increased the risks of harm from the research, or had an unfavorable impact on the risk/benefit ratio".
Arm/Group | Supervision/Paid/Open Group | Supervision/Paid/Closed Group | Supervision/Not Paid/Open Group | Supervision/Not Paid/Closed Group | Not Under Supervision/Paid/Open Group | Not Under Supervision/Paid/Closed Group | Not Under Supervision/Not Paid/Open Group | Not Under Supervision/Not Paid/Closed Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/20 | 0/25 | 0/22 | 0/32 | 0/22 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/20 | 0/25 | 0/22 | 0/32 | 0/22 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/20 | 0/25 | 0/22 | 2/32 | 0/22 | 0/15 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supervision/Paid/Open Group (N=15) | Supervision/Paid/Closed Group (N=20) | Supervision/Not Paid/Open Group (N=25) | Supervision/Not Paid/Closed Group (N=22) | Not Under Supervision/Paid/Open Group (N=32) | Not Under Supervision/Paid/Closed Group (N=22) | Not Under Supervision/Not Paid/Open Group (N=15) | Not Under Supervision/Not Paid/Closed Group (N=15)
Threat (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Participant reported receiving threats from a fellow participant via text message

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-01-29): https://cdn.clinicaltrials.gov/large-docs/91/NCT05934591/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT05934591/SAP_001.pdf
  • Informed Consent Form (2023-06-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT05934591/ICF_002.pdf